CLINICAL TRIAL: NCT01449136
Title: Phase 1 Study of Clinical and Radiographic Success of Antibacterial Cement in Infected Dentin of Deciduous Teeth
Brief Title: Use of Antibacterial Cement in Infected Dentin
Acronym: AC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Responsible Party: Principal Investigator, Jainara Maria Soares Ferreira, Principal investigator, University of Pernambuco
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1535/07
Record Dates: First submitted 2011-08-28; First posted 2011-10-10 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-09

CONDITIONS: Dental Caries
Keywords: Antibacterial agents; Deciduous Teeth; Clinical Trial
MeSH Terms: conditions — Dental Caries | interventions — Food, Formulated

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- antibacterial cement (Experimental)
  Interventions: Other: Antibacterial cement

INTERVENTIONS:
Other: Antibacterial cement — Glass ionomer cement containing 1% each of metronidazole, ciprofloxacin, and cefaclor
  Other Names: Antibacterial cement (Formula & Ação, São Paulo, Brazil)

SUMMARY:
Dental materials with antibacterial properties can prevent the harmful effects caused by oral cariogenic bacteria. This double-blind controlled clinical trial evaluated the performance of antibacterial cement for sealing infected dentin in atraumatic restorations of primary molars.

DETAILED DESCRIPTION:
The study enrolled 45 children (45 teeth) between 5 and 8 years of age, of both genders, divided into two groups. In group A (GA; n=22), the cavities were lined with conventional glass ionomer cement (Vidrion F®) and in group B (GB; n=23), with antibacterial cement (Vidrion F® containing 1% each of metronidazole, ciprofloxacin, and cefaclor). Both groups were restored with Ketac Molar Easymix®. Molars with carious lesions on the inner half of dentin without clinical or radiographic pulp damage were selected. Patients were evaluated clinically (for pain, fistulas, or mobility) and radiographically (area of caries, periapical region, and furcation of teeth) after 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* signed consent from a parent or guardian;
* primary molars with carious lesions on the inner half of dentin;
* access of caries lesions to dentin spoons.

Exclusion Criteria:

* damaged pulp determined clinically (for pain, fistulas, tooth mobility);
* damaged pulp determined radiography (bone or dental pathology);
* children taking antibiotics;
* children who refused the treatment;
* children had systemic disease.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
number of successful restorations with a dental liner with antibiotics | differences of overall success between baseline and the evaluations performed at 1, 3, 6, and 12 months.
  The absence of pain, fistulas, and mobility throughout the study was considered clinical success and the decreased or unchanged area of caries (obtained by a software to accurately measure distances between anatomical points selected by the operator of radiolucent zone beneath the restoration) and no bone or dental disorder was detected was considered radiographic success.
  Overall success was defined as clinical and radiographic success being achieved simultaneously.

CONTACTS AND LOCATIONS:
Locations (1):
- UFPB, João Pessoa, Paraíba, Brazil

REFERENCES:
- [Derived] Ferreira JM, Pinheiro SL, Sampaio FC, Menezes VA. Use of glass ionomer cement containing antibiotics to seal off infected dentin: a randomized clinical trial. Braz Dent J. 2013;24(1):68-73. doi: 10.1590/0103-6440201301925. PMID 23657417